CLINICAL TRIAL: NCT05376137
Title: Personal Therapy Comfort Settings Pilot Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA11022022
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Default comfort settings (Active Comparator): Comfort settings will be set to default (out of the box setttings)
  Interventions: Device: continuous positive airway pressure (CPAP)
- Personalized Therapy Comfort Settings (Experimental): Comfort settings will be personalized to each user
  Interventions: Device: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: continuous positive airway pressure (CPAP) — CPAP comfort settings will be modified in the active group to be personalized to each participant

SUMMARY:
350 participants will be enrolled in this study. The target population are patients newly diagnosed with OSA and starting CPAP treatment.

User accessible customizable comfort settings (Response setting, expiratory pressure relief (EPR) on/off and EPR level, and Ramp) will be set to either default (control group), or personalized for that participant (active treatment group).

Usage will be recorded for the first 1 month of CPAP treatment, to determine if customizing comfort settings can improve CPAP compliance

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients who are ≥ 18 years of age
* Patients newly diagnosed with OSA and indicated for CPAP therapy.

Exclusion Criteria:

* Patients who have previously used PAP therapy
* Patients who require a bilevel device
* Patients who are or may be pregnant

  * Patients who are unable to attend follow up appointments
* Patients with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury
* Patients believed to be unsuitable for inclusion by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Comparison of treatment continuance between the control group and active treatment group. | 4 weeks after commencement of CPAP
  Patients who drop off treatment (stop using CPAP treatment) in each group will be compared after 1.5 months of CPAP treatment.

SECONDARY OUTCOMES:
comparison of compliance between the control group and active treatment group | 4 weeks after commencement of CPAP
  Usage will be compared between the two groups
Treatment efficacy | 4 weeks after commencement of CPAP
  Residual Apnea-hypopnea index will be compared between the two groups
Mask leak | 4 weeks after commencement of CPAP
  Mask leak will be compared between the two groups
Settings changes | 4 weeks after commencement of CPAP
  Number of comfort settings changes will be compared between the two groups
Ad hoc contacts | 4 weeks after commencement of CPAP
  Number of ad hoc contacts between participants and clinicians will be compared between the two groups

OTHER OUTCOMES:
Exploratory analysis of long term usage | 3,6,9, 12 months after commencement of CPAP
  CPAP usage will be compared at 3, 6, 9 and 12 months for patients who have consented, as an exploratory analysis of long term usage

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Armitstead, PhD, Principal Investigator — ResMed
Locations (1):
- ResMed Centre for Healthy Sleep, Bella Vista, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No